CLINICAL TRIAL: NCT05832034
Title: Treatment With add-on IVIg in Myositis Early In the diSease Course May be sUperior to Steroids Alone for Reaching CLinical improvemEnt
Brief Title: Add-on Intravenous Immunoglobulins in Early Myositis
Acronym: TIMEISMUSCLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Princess Beatrix Muscle Foundation (Other)
Responsible Party: Principal Investigator, Joost Raaphorst, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL74270.018.20
Record Dates: First submitted 2022-02-21; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Inflammatory Myopathy, Idiopathic; Dermatomyositis; Antisynthetase Syndrome; Immune-Mediated Necrotizing Myopathy; Polymyositis; Myositis
Keywords: Myositis; Inflammatory myopathies; Intravenous immunoglobulins; Early symptomatic
MeSH Terms: conditions — Myositis; Dermatomyositis; Antisynthetase syndrome; Polymyositis | interventions — Immunoglobulins, Intravenous; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Home-care nurse preparing study medication will be unblinded. Home-care nurse is not involved in outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Add-on IVIg (Experimental): Patients in the intervention arm will be treated with Nanogam® in a dosage of 2 g/kg over 2-5 days, with a maximum of 80 g/day and a total of 180 gram at baseline and after 4 and 8 weeks. Nanogam® contains 100 mg/mL normal human immunoglobulin with a purity of at least 95% IgG and a maximum of 12 microgram/mL IgA, in a solution of water for injections and glucose. The first 30 grams are administered in hospital.
  Interventions: Drug: Immune Globulin Intravenous (Human)
- Placebo (Placebo Comparator): Patients in the control arm will be treated with placebo infusions, containing sodium chloride 0.9%, at baseline and after 4 and 8 weeks. The first 30 grams are administered at the neurology ward, after 4 and 8 weeks infusions will be administered at home
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Immune Globulin Intravenous (Human) — IVIg is 2 g/kg over 2 to 5 days at baseline, followed by 2 g/kg IV in 2 to 5 days after 4 and 8 weeks. The rate of infusion is controlled by means of an infusion pump. The first dosage (30 grams IVIg) will be administered on the neurology ward.
  Other Names: Nanogam
  Arms: Add-on IVIg
Drug: Placebo — Placebo infusions, containing sodium chloride 0.9%, at baseline and after 4 and 8 weeks.
  Other Names: Sodium chloride or saline 0.9%
  Arms: Placebo

SUMMARY:
In patients with myositis early immunomodulation by intensive treatment ("hit-early/hit-hard" principle) may induce faster reduction of disease activity and prevent chronic disability. Intravenous immunoglobulin (IVIg) in addition to standard treatment with glucocorticoids may be beneficial for this purpose: add-on IVIg improved symptoms in steroid-resistant myositis, and first-line monotherapy IVIg led to a fast and clinically relevant response in a pilot study in nearly 50% of patients with myositis.

DETAILED DESCRIPTION:
Considering the known effects of IVIg in idiopathic inflammatory myopathies (IIM), both as add-on therapy in refractory patients, as well as monotherapy in newly diagnosed IIM, we conducted a phase-2 double-blind placebo-controlled randomized trial to investigate the effect of add-on IVIg in patients with newly diagnosed IIM, who are treated with monotherapy prednisone.

Objective:

The primary aim of this trial is to examine whether the addition of early administered IVIg to standard therapy with prednisone in patients with newly diagnosed myositis leads to an improved clinical response after 12 weeks, compared to prednisone and placebo. Clinical response will be measured as the difference of the mean TIS after 12 weeks between intervention and control groups.

The secondary aims are to examine whether the intervention leads to a shorter time to improvement, and sustained positive effects on health-related quality of life, physical activity and fatigue, and a sustained reduction of muscle MRI abnormalities, as assessed up to 52 weeks.

Following a screening visit at the outpatient clinic, patients will be admitted to the neurology ward of the Amsterdam University Medical Center (AUMC) for the first infusion of study treatment. The remaining study medication will be administered at home, according to routine clinical practice for IVIg treatment in neuromuscular disorders in the Netherlands. A second and third study treatment will be administered at home after 4 and 8 weeks. At baseline and after 4, 8, 12, 26 and 52 weeks outcome assessments will be performed at the outpatient clinic. The outpatient study clinic visits at baseline and after 4, 12, 26 and 52 weeks will be combined with regular outpatient clinic visits.

The additional burden related to outcome assessments will consist of MRI muscle imaging after 12 weeks, blood sampling after 2, 4, 6, and 10 weeks and filling in questionnaires at baseline and after 4, 8, 12, 26 and 52 weeks. In addition, participants are asked to wear a watch three times in a period of 12 weeks and after 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with IIM, according to diagnostic criteria:

  * Dermatomyositis
  * Polymyositis
  * Anti-synthetase syndrome
  * Immune mediated necrotizing myopathy
  * Overlap myositis
* Disease duration < 12 months
* Minimal disability defined as at least 10% loss on Manual Muscle Testing (MMT) and abnormal scores on two other Core Set Measures (CSMs) of the international Myositis Assessment and Clinical Studies (IMACS) group (see 'Primary and secondary outcomes').
* Patients are eligible for inclusion if they are treatment-naive, or if there is no clinical evident response (as carefully judged by the treating physician at a screening visit) to prior treatment with:
* High dosed glucocorticoids, such as dexamethasone (e.g. 40 mg per day up to 4 days) or intravenous methylprednisolone (e.g. 1000 mg daily for three days), within 1 week prior to screening visit.
* Daily dosed prednisone 1 mg/kg, or equivalent, used for up to 2 weeks prior to screening visit.
* Treatment with low-dosed prednisone (max 20 mg daily) up to three months prior to screening visit.
* Treatment with biologicals or other immunosuppressive or immunomodulatory treatment when meeting all of the following criteria:

  * Stable dose for the last 6 months
  * The biological or other immunosuppressive or immunomodulatory treatment has been approved for a non-muscular condition (e.g. hematological condition, eczema) and is not known for its use in idiopathic inflammatory myopathy
  * The biological or other immunosuppressive or immunomodulatory treatment is not known to induce inflammatory myopathy
* Signed informed consent

Exclusion Criteria:

A potentially eligible patient who meets any of the following criteria will be excluded from participation in this study:

* Severe muscle weakness (i.e. bedridden, severe dysphagia requiring a feeding tube, or respiratory muscle weakness (forced vital capacity below 50% of predicted in upright position)) necessitating more intensive treatment than standard glucocorticoids from the start.
* Related to IVIg:

  * History of thrombotic episodes within 10 years prior to enrolment
  * Known allergic reactions or other severe reactions to any blood-derived product
  * Known Immunoglobulin A (IgA) deficiency and IgA serum antibodies
  * Pregnancy or trying to conceive
  * Use of loop diuretics
  * Use of nephrotoxic medication
* Conditions that are likely to interfere with:

  * Compliance (legally incompetent and/or incapacitated patients are excluded), or,
  * Evaluation of efficacy (e.g. due to severe pre-existing disability as a result of any other disease than myositis or due to language barrier)
* Immunosuppressive medication or immunomodulatory treatment within the last 3 months (e.g. azathioprine, methotrexate, mycophenolate mofetil, tacrolimus, cyclophosphamide, cyclosporine, IVIg, biologicals, Janus kinase inhibitors, plasmapheresis).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in Total Improvement Score (TIS) | Baseline and week 12
  The primary outcome is the Total Improvement Score (TIS) of the myositis response criteria after 12 weeks, measured as the difference of the mean TIS after 12 weeks between intervention and control groups. Total Improvement Score (TIS) is based on 6 validated core set measures (CSMs), which each determine disease activity as defined by the International Myositis Assessment and Clinical Studies (IMACS) group. TIS ranges between 0 and 100 and corresponds to a degree of improvement; higher scores correspond to a greater degree of improvement.

SECONDARY OUTCOMES:
Time to response (TIS>40 points) | Will be examined at week 4, 8, 12, 26 and 52 weeks.
  This is defined as the time is taken to reach a Total Improvement Score > 40 points.Total Improvement Score is based on 6 validated core set measures (CSMs), which each determine disease activity as defined by the International Myositis Assessment and Clinical Studies (IMACS) group.
Total Improvement Score (IMACS). | TIS will be assessed at t = 0, and after 4, 8, 12, 26 and 52 weeks
  Total Improvement Score (TIS) is based on 6 validated core set measures (CSMs), which each determine disease activity as defined by the International Myositis Assessment and Clinical Studies (IMACS) group. TIS ranges between 0 and 100 and corresponds to a degree of improvement; higher scores correspond to a greater degree of improvement.
Core set measures (CSM) - physician global activity (PhGA) | CSMs will be assessed at baseline, week 4, 8, 12, 26 and 52.
  1. physician global activity (PhGA): assessment of global disease activity on a 10 cm Visual Analogue Scale (VAS) by the treating physician. 0 = no disease activity, 10 most activity
  On a total of 6 CSM
Core set measures (CSM) - patient global activity (PGA) | CSMs will be assessed at baseline, week 4, 8, 12, 26 and 52.
  2. patient global activity (PGA): assessment of global disease activity on a 10 cm VAS by the patient. 0 = no disease activity, 10 most activity On a total of 6 CSM
Core set measures (CSM) - Manual Muscle Testing (MMT) | CSMs will be assessed at baseline, week 4, 8, 12, 26 and 52.
  3. Manual Muscle Testing (MMT): sum score of 12 proximal+distal and 2 axial muscle groups. Score 0 - 260 (no muscle weakness). 0 = zero contractions in muscle, 10 = normal On a total of 6 CSM
Core set measures (CSM) - Health Assessment Questionnaire (HAQ) | CSMs will be assessed at baseline, week 4, 8, 12, 26 and 52.
  4. Health Assessment Questionnaire (HAQ): average of a survey scoring 8 domains, from 0 (without any difficulty) to 3 (unable to do) On a total of 6 CSM
Core set measures (CSM) - Serum muscle enzyme activities | CSMs will be assessed at baseline, week 4, 8, 12, 26 and 52.
  5. Serum muscle enzyme activities expressed as the most abnormal one in the upper limit of normal.
  On a total of 6 CSM
Core set measures (CSM) - Extramuscular disease activity | CSMs will be assessed at baseline, week 4, 8, 12, 26 and 52.
  6. Extramuscular disease activity on a 10 cm VAS based on the Myositis Disease Activity Assessment, measuring the degree of disease activity of extra-muscular organ systems. Score is based on a 0 - 4 scale, related to worsening or improvement.
  On a total of 6 CSM
Patient-Reported Outcome Measures (PROMs) questionnaire - Fatigue | At baseline, and after 4, 8, 12, 26 and 52 weeks.
  These PROMs relate to different aspects of quality of life, this questionnaire specified on fatigue. The three PROMs are offered as Short Forms: fixed set of 4-10 questions for one of each domain.
  Each item is scored on a 5-point Likert scale, with higher scores indicating better functioning, and item category responses range from 1 to 5.
  For example: 1= not at al, 2 = a little, 3 = moderately, 4 = mostly, 5= completely.
Patient-Reported Outcome Measures (PROMs) questionnaire - Pain interference | At baseline, and after 4, 8, 12, 26 and 52 weeks.
  These PROMs relate to different aspects of quality of life, this questionnaire specified on pain interference (in life). The three PROMs are offered as Short Forms: fixed set of 4-10 questions for one of each domain.
  Each item is scored on a 5-point Likert scale, with higher scores indicating better functioning, and item category responses range from 1 to 5.
  For example: 1= not at al, 2 = a little, 3 = moderately, 4 = mostly, 5= completely.
Patient-Reported Outcome Measures (PROMs) questionnaire - Physical function | At baseline, and after 4, 8, 12, 26 and 52 weeks.
  These PROMs relate to different aspects of quality of life, this questionnaire specified on physical function. The three PROMs are offered as Short Forms: fixed set of 4-10 questions for one of each domain.
  Each item is scored on a 5-point Likert scale, with higher scores indicating better functioning, and item category responses range from 1 to 5.
  For example: 1= not at al, 2 = a little, 3 = moderately, 4 = mostly, 5= completely.
Fatigue | At baseline, and after 4, 8, 12, 26 and 52 weeks.
  The second most important domain according to patients with myositis and health-care providers (OMERACT study group). We will use the Checklist Individual Strength (CIS)-fatigue, a generic fatigue scale, which has been validated in neuromuscular disorders.
Health related quality of life (HR-QoL) | At baseline, and after 4, 8, 12, 26 and 52 weeks.
  HR-QoL will be assessed with EuroQol Group Health Questionnaire (EQ5D). EQ5D is a widely used questionnaire for assessment of general health and has shown responsivity in our previous study on monotherapy IVIg in IIM
Physical activity | Two consecutive weeks, at baseline, week 4, week 8 and week 26.
  Accelerometry will be used to measure physical activity, patients will be offered a wrist-worn wearable (Actigraph GT9X32). For accelerometry we will calculate the mean number of steps and the mean number of flights of stairs per 24 hours, during the 5 most active days per week.
Mean daily prednisone dosage | Calculated at week 4, 8, 12, 26 and 52.
  Start dosage 1 mg/kg (maximum 80 mg). A standard tapering scheme in the first months consists of 10 mg reduction of dosage every 4 weeks.
Muscle hyperintensities. | At baseline, and after 12 and 26 weeks.
  Indicative for edema (T2/STIR) and fatty infiltration (T1) on total body MRI. The MRI results will be used as a marker of inflammation and disease damage, respectively. Sum scores of semi-quantitatively rated muscle edema and fatty infiltration will be calculated. For this parameters we will examine the interaction between time and group.
IgG blood levels. | Obtained immediately before, and two weeks after the administration of study medication
  Immunoglobulin G (IgG) levels in serum samples will be measured by turbidimetry.
Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI). | At baseline, and after 4, 8, 12, 26 and 52 weeks.
  In the subgroup of patients with dermatomyositis, this validated tool will be used to characterize cutaneous dermatomyositis severity and detect improvement in disease activity.
Composite questionnaire on health care use and productivity loss. | At baseline and week 12
  This questionnaire is based on the Medical Consumption Questionnaire (iMCQ) and the Productivity Cost Questionnaire (iPCQ) and is currently being used in the OPTIC trial (add-on prednisone in chronic inflammatory demyelinating polyneuropathy (CIDP)).

CONTACTS AND LOCATIONS:
Overall Officials: Raaphorst, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Department of Neurology, Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oddis CV, Aggarwal R. Treatment in myositis. Nat Rev Rheumatol. 2018 May;14(5):279-289. doi: 10.1038/nrrheum.2018.42. Epub 2018 Mar 29. PMID 29593343
- [Background] Aggarwal R, Rider LG, Ruperto N, Bayat N, Erman B, Feldman BM, Oddis CV, Amato AA, Chinoy H, Cooper RG, Dastmalchi M, Fiorentino D, Isenberg D, Katz JD, Mammen A, de Visser M, Ytterberg SR, Lundberg IE, Chung L, Danko K, Garcia-De la Torre I, Song YW, Villa L, Rinaldi M, Rockette H, Lachenbruch PA, Miller FW, Vencovsky J; International Myositis Assessment and Clinical Studies Group and the Paediatric Rheumatology International Trials Organisation. 2016 American College of Rheumatology/European League Against Rheumatism criteria for minimal, moderate, and major clinical response in adult dermatomyositis and polymyositis: An International Myositis Assessment and Clinical Studies Group/Paediatric Rheumatology International Trials Organisation Collaborative Initiative. Ann Rheum Dis. 2017 May;76(5):792-801. doi: 10.1136/annrheumdis-2017-211400. PMID 28385805
- [Background] Hoogendijk JE, Amato AA, Lecky BR, Choy EH, Lundberg IE, Rose MR, Vencovsky J, de Visser M, Hughes RA. 119th ENMC international workshop: trial design in adult idiopathic inflammatory myopathies, with the exception of inclusion body myositis, 10-12 October 2003, Naarden, The Netherlands. Neuromuscul Disord. 2004 May;14(5):337-45. doi: 10.1016/j.nmd.2004.02.006. No abstract available. PMID 15099594
- [Background] Dalakas MC, Illa I, Dambrosia JM, Soueidan SA, Stein DP, Otero C, Dinsmore ST, McCrosky S. A controlled trial of high-dose intravenous immune globulin infusions as treatment for dermatomyositis. N Engl J Med. 1993 Dec 30;329(27):1993-2000. doi: 10.1056/NEJM199312303292704. PMID 8247075
- [Background] Mecoli CA, Park JK, Alexanderson H, Regardt M, Needham M, de Groot I, Sarver C, Lundberg IE, Shea B, de Visser M, Song YW, Bingham CO 3rd, Christopher-Stine L. Perceptions of Patients, Caregivers, and Healthcare Providers of Idiopathic Inflammatory Myopathies: An International OMERACT Study. J Rheumatol. 2019 Jan;46(1):106-111. doi: 10.3899/jrheum.180353. Epub 2018 Sep 15. PMID 30219767
- [Background] Malattia C, Damasio MB, Madeo A, Pistorio A, Providenti A, Pederzoli S, Viola S, Buoncompagni A, Mattiuz C, Beltramo A, Consolaro A, Ravelli A, Ruperto N, Picco P, Magnano GM, Martini A. Whole-body MRI in the assessment of disease activity in juvenile dermatomyositis. Ann Rheum Dis. 2014 Jun;73(6):1083-90. doi: 10.1136/annrheumdis-2012-202915. Epub 2013 May 1. PMID 23636654
- [Background] Lim J, Eftimov F, Verhamme C, Brusse E, Hoogendijk JE, Saris CGJ, Raaphorst J, De Haan RJ, van Schaik IN, Aronica E, de Visser M, van der Kooi AJ. Intravenous immunoglobulins as first-line treatment in idiopathic inflammatory myopathies: a pilot study. Rheumatology (Oxford). 2021 Apr 6;60(4):1784-1792. doi: 10.1093/rheumatology/keaa459. PMID 33099648